CLINICAL TRIAL: NCT07367932
Title: Crisaborole 2% Versus Tacrolimus 0.03% Ointments for the Treatment of Mild to Moderate Atopic Dermatitis: A Comparative Study
Brief Title: Comparative Study of Crisaborole vs. Tacrolimus in Atopic Dermatitis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Elbendary, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS-61-2025
Record Dates: First submitted 2025-12-28; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Dermatitis, Atopic; Eczema
Keywords: Tacrolimus; Crisaborole; Atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crisaborole ointment (Active Comparator)
  Interventions: Drug: Application of crisaborole twice daily
- Tacrolimus ointment (Active Comparator)
  Interventions: Drug: Tacrolimus ointment in atopic dermatitis

INTERVENTIONS:
Drug: Application of crisaborole twice daily — compare the efficacy and safety of crisaborole ointment on mild to moderate atopic dermatitis for 1 month and followup in 2 months
  Arms: Crisaborole ointment
Drug: Tacrolimus ointment in atopic dermatitis — compare the efficacy and safety of tacrolimus ointment, in the treatment of patients with mild-to-moderate atopic dermatitis
  Arms: Tacrolimus ointment

SUMMARY:
This study will compare the efficacy and safety of crisaborole ointment with tacrolimus ointment, in the treatment of patients with mild-to-moderate atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of AD, according to Hanifin and Rajka criteria.
* Patients of both genders
* Age 5-25 years
* Baseline Investigator's Static Global Assessment (ISGA) score of mild (2) or moderate (3).

Exclusion Criteria:

* Clinically infected eczema.
* Baseline Investigator's Static Global Assessment (ISGA) score of severe (4).
* Associated comorbidities that exacerbate pruritus.
* Patients receiving topical treatment for AD and/or pruritus within the past 14 days and/or systemic treatment within the past month.
* Pregnancy and lactation if in the childbearing period

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Improvement of Investigator's Static Global Assessment score | 3 months
  1. Assessment of the **Investigator's Static Global Assessment** scores before and after treatment with crisaborole 2% ointment.
  2. Assessment of the **Investigator's Static Global Assessment** before and after treatment with tacrolimus 0.03% ointment.
  3. Comparison of the **percentage of improvement** in the **Investigator's Static Global Assessment** between the two treatment groups.
Improvement of Eczema Area and Severity Index | 3 months
  1. Assessment of **Eczema Area and Severity Index** scores before and after the use of **crisaborole 2% ointment**.
  2. Assessment of **Eczema Area and Severity Index** scores before and after the use of **tacrolimus 0.03% ointment**.
  3. Comparison of the percentage of improvement in the **Eczema Area and Severity Index** scores between the two treatment groups